CLINICAL TRIAL: NCT02551380
Title: Evaluation of the Efficiency of Folinic Acid in Children With Autism Spectrum Disorders: a Pilot Study "EFFET"
Brief Title: Folinic Acid in Children With Autism Spectrum Disorders
Acronym: EFFET
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015-000955-25
Record Dates: First submitted 2015-09-14; First posted 2015-09-16 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Leucovorin; Lactose

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treated (Experimental): treatment with Folinoral (folinic acid) 5mg twice a day (10 mg per day) during 12 weeks
  Interventions: Drug: FOLINORAL
- control (Placebo Comparator): treatment with one capsule of placebo twice a day during 12 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: FOLINORAL — Folinoral (folinic acid) 5mg twice a day (10 mg per day) during 12 weeks
  Other Names: Folinic acid
  Arms: Treated
Other: Placebo — Placebo 5mg twice a day (10 mg per day) during 12 weeks
  Other Names: Lactose
  Arms: control

SUMMARY:
The investigator planned to study the efficiency of folinic acid treatment on autistic symptoms in children suffering from autism spectrum disorder.

DETAILED DESCRIPTION:
The aim of this study is to realise a pilot study in France in order to evaluate the efficiency of folinic acid in treatment of autism spectrum disorder and get first estimations about prevalence of auto antibodies anti-FRα in France.

The study is a randomized controlled trial monocentric,evaluating folinic acid 10mg per day versus placebo, in single-blind during 12 weeks.

Primary objective : The primary objective is to evaluate the efficiency of folinic acid (calcium folinate) 5mg twice a day during 12 weeks on reduction of autistic troubles, particularly on communication and social interaction

Secondary objective :

* Evaluate the efficiency of folinic acid on reduction of autistic symptoms perceived by parents
* Evaluate the constancy of auto antibodies anti-FRα rates

ELIGIBILITY:
Inclusion Criteria:

1. Children with autism spectrum disorders defined by : Autism Diagnostic Observation Schedule (ADOS), Autism Diagnostic Interview (ADI), Childhood Autism Rating Scale (CARS) or diagnosed by a physician (pediatrician, child psychiatrist)
2. Children aged 3 to 10 years
3. Weight> 10 kg
4. Language impairment (based on the medical assessment)
5. Ability to maintain other therapies started before the study
6. No changes of therapeutic treatments within the 8 weeks before the start of the study

Exclusion Criteria:

1. Treatment may impair folate metabolism (methotrexate, anticonvulsivants : phenobarbital sodium valproate, phenytoin, primidone, carbamazepine, valproic acid, divalproex, antibiotics : tetracycline, trimethoprim, pyrimethamine, inhibitors of proton pump inhibitors of histamine-2)
2. Antipsychotic treatment (including treatment with Risperidone)
3. Vitamin or mineral supplementation exceeding guidelines
4. Children with severe irritability (Aberrant Behavior Checklist> 17)
5. Gastroesophageal reflux disease
6. Any known renal or liver disease
7. Child born premature (<37SA)
8. Known intolerance to lactose
9. Hypersensitivity / allergic reaction to calcium folinate
10. The sibling children with autism spectrum disorders

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2015-10; Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of severity of autistic symptoms with standardized scale ADOS (Autism Diagnosis Observation Scale) | change in ADOS scale at 12 weeks
  Autistic symptoms (particularly communication and social interaction) measured by standardized scale ADOS (Autism Diagnosis Observation Scale) : comparison of score between folinic acid group and placebo at T0 et after 12 weeks of treatment

SECONDARY OUTCOMES:
Evaluation of the reduction of autistic symptom perceived by parents with a heteroevaluation scale : SRS (social responsiveness scale) | Change in SRS at 12 weeks
  - Evaluation of the reduction of autistic symptom perceived by parents with a heteroevaluation scale : SRS (social responsiveness scale)
  o Comparison of score between folinic acid group and placebo group at T0 (inclusion) and after 12 weeks of treatment
evaluate the constancy of auto antibodies anti-FRα | change of auto antibodies anti-FRα at 12 weeks
  Serum dosage of auto antibodies anti-FRα at T0 and at 12 weeks to evaluate the constancy of auto antibodies anti-FRα

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Leheup, M.D, Ph.D, Principal Investigator — CHU NANCY- Hopital Brabois Enfants
Locations (1):
- CHU Nancy-Hopital Brabois Enfants, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: Undecided
To be completed after discussions with the different research teams participating in the study